CLINICAL TRIAL: NCT02853708
Title: Epidemiology of ST131 in Besançon University Hospital
Acronym: coliST131
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2015/62
Record Dates: First submitted 2016-07-19; First posted 2016-08-03 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Escherichia Coli Infections
Keywords: E. coli; extended-spectrum beta-lactamase; molecular epidemiology; risk factors
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial isolate
Oversight: Data Monitoring Committee: No

SUMMARY:
The sequence type 131 (ST131) is a predominant lineage among extraintestinal pathogenic Escherichia coli. It plays a major role in the worldwide dissemination of E. coli that produce extended-spectrum beta-lactamase (ESBL). The aim of this study was to describe the epidemiology of ESBL producing ST131clonal group in our university hospital. All patients with an infection due to ESBL E. coli will be prospectively included for a 2-year period. ST131 isolates will be identified and risk factors associated to ST131 will be determined in comparison to non-ST131 ESBL E. coli.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with ESBL producing E. coli

Exclusion Criteria:

* Patients known to be carrier or infected in the previous year, patients only colonised with ESBL producing E. coli.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized at CHRU Besançon and infected with ESBL producing E. coli
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Risk factors associated to ESBL ST 131 infections | up to 2 years
  Time of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicolas-Chanoine MH, Bertrand X, Madec JY. Escherichia coli ST131, an intriguing clonal group. Clin Microbiol Rev. 2014 Jul;27(3):543-74. doi: 10.1128/CMR.00125-13. PMID 24982321
- [Background] Lafolie J, Nicolas-Chanoine MH, Grenouillet F, Hocquet D, Bertrand X. Prevalence of Escherichia coli sequence type 131 and its H30 subclone among E. coli isolates in a French hospital. Int J Antimicrob Agents. 2014 Nov;44(5):466-8. doi: 10.1016/j.ijantimicag.2014.07.016. Epub 2014 Sep 3. PMID 25241262
- [Background] Lafolie J, Sauget M, Cabrolier N, Hocquet D, Bertrand X. Detection of Escherichia coli sequence type 131 by matrix-assisted laser desorption ionization time-of-flight mass spectrometry: implications for infection control policies? J Hosp Infect. 2015 Jul;90(3):208-12. doi: 10.1016/j.jhin.2014.12.022. Epub 2015 Feb 28. PMID 25799482
- [Background] Can F, Azap OK, Seref C, Ispir P, Arslan H, Ergonul O. Emerging Escherichia coli O25b/ST131 clone predicts treatment failure in urinary tract infections. Clin Infect Dis. 2015 Feb 15;60(4):523-7. doi: 10.1093/cid/ciu864. Epub 2014 Nov 6. PMID 25378460